CLINICAL TRIAL: NCT06274177
Title: Evaluation of the Safety and Efficacy of the BTL-785F Device for Non-invasive Submental Fat Reduction and Neck Rejuvenation
Brief Title: Evaluation of the BTL-785F Device for Submental Fat Reduction and Neck Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-785_CTUS1400
Record Dates: First submitted 2024-02-07; First posted 2024-02-23 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Fat Burn
Keywords: submentum; neck rejuvenation; double chin; fat
MeSH Terms: conditions — Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with BTL-785-7 (Experimental): Treatment with BTL-785F device (BTL-785-7 applicator)
  Interventions: Device: BTL-785-7

INTERVENTIONS:
Device: BTL-785-7 — Treatment with the BTL-785F device with the BTL-785-7 applicator for non-invasive reduction of submental fat and skin laxity treatment

SUMMARY:
This study will evaluate the clinical safety and the performance of the BTL-785F system equipped with the BTL-785-7 applicator for non-invasive reduction of submental fat and skin laxity treatment.

DETAILED DESCRIPTION:
This is a multi center single-arm, open-label, interventional study.

The subjects will be enrolled and assigned into one experimental study arm. The subjects will be required to complete four (4) treatment visits and two follow-up visits.

At baseline inclusion and exclusion criteria will be verified upon obtaining informed consent from the patient.

The treatment administration phase consists of four (4) treatment visits, delivered 5-10 days apart. Follow-ups visits at 1 month and 3 months after the final treatment will be held.

At every treatment visit after the first, prior to the procedure, the participants will be assessed for adverse effects resulting from the previous treatment(s) with the BTL-785F device.

Safety measures will include documentation of adverse events (AE) during and after the procedures and if needed medical assistance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 21 years of age seeking treatment for reduction of submental fat
* Subjects should be able understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form
* Presence of clearly visible excess fat in submentum as deemed appropriate by the Investigator
* Subjects willing and able to abstain from partaking in any facial treatments other than the study procedure during study participation
* Willingness to comply with study instructions, to return to the clinic for the required visits, and to have photographs of their face taken

Exclusion Criteria:

* Local bacterial or viral infection in the area to be treated
* Local acute inflammation in the area to be treated
* Impaired immune system caused by any immunosuppressive illness, disease or medication
* Isotretinoin and tretinoin-containing medication use in the past 12 months
* Skin related autoimmune diseases
* Radiation therapy and/or chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Facial dermabrasion, facial resurfacing, or deep chemical peeling in the treatment area within 3 months prior to the treatment
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of skin disorders, keloids, abnormal wound healing and dry or fragile skin
* History of any type of cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis, hypersensitive carotid sinus and thrombosis)1
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Acute neuralgia and neuropathy
* Kidney or liver failure
* Nerve insensitivity (sensitivity disorders) to heat in the treatment area
* Varicose veins, pronounced edemas1
* Prior use of dermal fillers, botulinum toxin, lasers, etc. therapies in the treated area that can influence the study results at the investigator discretion
* Unwillingness/inability to not change their usual cosmetics and especially not to use fat reduction, anti-aging or anti-wrinkles products in the treated area during the duration of the study including the follow-up period
* Electroanalgesia without exact diagnosis of pain etiology
* Neurological disorders (such as multiple cerebrospinal sclerosis, epilepsy)
* Blood vessels and lymphatic vessels inflammation
* Any other disease or condition at the investigator discretion that may pose risk to the patient or compromise the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2024-08-04 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Submental fat thickness reduction | 15 months
  The primary efficacy outcome measure is a statistically significant reduction of at least 1.0 mm in the average submental fat layer thickness in the majority of subjects measured by MRI at 3-months follow-up compared to baseline.

SECONDARY OUTCOMES:
Incidence of Treatment-related Adverse Events | 15 months
  To evaluate the safety of the BTL-785F device with the BTL-785-7 applicator for non-invasive reduction of submental fat through monitoring of adverse reactions.
Change on the Clinician Reported - Submental Fat Rating Scale score | 15 months
  Evaluation of the change in the Clinician Reported - Submental Fat Rating Scale (CR-SMFRS) grade. The scale ranges from grade 0 (no evident submental fat) to grade 4 (extreme submental convexity). Photographs from the last therapy, 1 month and 3 months follow-up will be compared to baseline photographs. An improvement is considered a decrease of the grade in the Clinician Reported - Submental Fat Rating Scale.
Satisfaction Assessed by the Satisfaction Questionnaire | 15 months
  The 5-point Likert scale Subject Satisfaction Questionnaire will be used for evaluating the satisfaction. The Subject Satisfaction Questionnaire will be given to subjects after the last therapy, at 1-month and 3-month follow-up. The answers to the questions related to the subjects' under-chin and overall facial appearance will vary from "strongly agree" to "strongly disagree".
Change in the submental-cervical angle | 15 months
  Statistically significant change in submental-cervical angle (SCA) convexity in the majority of the subjects
Comfort Assessed by Therapy Comfort Questionnaire | 15 months
  The 5-point Likert scale Therapy Comfort questionnaire will be used for evaluating the comfort during the treatment sessions. Pain sensation will be rated by the subjects from 0 (no pain) to 10 (worst possible pain). The Therapy Comfort questionnaire will be given to subjects after the last therapy.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Precision Skin LLC, Davie, Florida
  - Chicago Cosmetic and Dermatologic Research, Chicago, Illinois
  - New Jersey Plastic Surgery (NJPS), Montclair, New Jersey
  - Gentile Facial Plastic and Aesthetic Laser Center, Youngstown, Ohio

IPD SHARING:
Plan to Share IPD: No